CLINICAL TRIAL: NCT01313819
Title: A Double Blind, Placebo-controlled Study for the Effect of IV Amantadine on Freezing of Gait (FOG) Resistant to Dopaminergic Therapy
Brief Title: The Effect of IV Amantadine on Freezing of Gait (FOG) Resistant to Dopaminergic Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, BS Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H-1012-044-344
Record Dates: First submitted 2011-03-10; First posted 2011-03-14 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Parkinson's Disease; Freezing of Gait
Keywords: Freezing
MeSH Terms: conditions — Parkinson Disease | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Give IV amantadine first then IV placebo(normal saline) drug
  Interventions: Drug: PK-Merz® 200mg/500ml inj(Amantadine) , Normal saline 500ml inj
- Group 2 (Active Comparator): Give IV placebo drug first then IV amantadine
  Interventions: Drug: PK-Merz® 200mg/500ml inj(Amantadine) , Normal saline 500ml inj

INTERVENTIONS:
Drug: PK-Merz® 200mg/500ml inj(Amantadine) , Normal saline 500ml inj — IV amantadine at 200 mg in 500 cm3 of saline solution or normal saline 500 cm3 given over a 3-h period, twice a day for 2 days along with the pre-existing dopaminergic and non-dopaminergic medication

SUMMARY:
Tp determine the effect of IV amantadine on dopaminergic-drug-resistant freezing of gait(FOG)in patients with Parkinson's disease

DETAILED DESCRIPTION:
1. Freezing of gait (FOG) is one of the most disabling symptoms of Parkinson's disease.

   We experienced that severe FOG was markedly improved by IV amantadine in the patients who had Parkinson's disease. But IV drug may have placebo effect. Therefore, We designed double blind, placebo controlled study to know whether IV amantadine is effective in the patient with dopaminergic-drug-resistant freezing of gait(FOG).
2. Cross over study design

   * Compare the change of FOGQ(freezing of gait questionaire) score from the baseline to IV amantadine and placebo drug
   * randomized assigned order of amantadine and placebo drug.
   * investigator of FOG: blinded to the order of drugs
   * each patient has IV drug for 2 days for each drug

ELIGIBILITY:
Inclusion Criteria

* age: 30-80 years
* idiopathic Parkinson's disease
* The patient must be taking optimised levodopa/DDI therapy (based on investigator's judgement) during OPD observation period, though the patient have FOG-Q score ≥ 10 points even though On-state.

Exclusion Criteria:

* "Off" freezing:The patient has improved FOG in "On" state
* clinically significant or unstable medical or surgical condition
* The patient has Parkinson plus like MSA, PSP, and PPFG, and secondary parkinsonism like NPH, vascular parkinsonism, postencephalitic parkinsonism, CO poisoning.
* history of seizure.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
change of FOGQ score | 2 days for each drug

SECONDARY OUTCOMES:
UPDRS and HY stage | 2 days for each drug
side effect | 2 days, 2 weeks after discharge
Patient global impression | 2 days, 2 weeks after discharge
4*10m walk test | 2 days for each drug

CONTACTS AND LOCATIONS:
Overall Officials: Beom S Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Giladi N, Kao R, Fahn S. Freezing phenomenon in patients with parkinsonian syndromes. Mov Disord. 1997 May;12(3):302-5. doi: 10.1002/mds.870120307. PMID 9159723
- [Background] Giladi N. Medical treatment of freezing of gait. Mov Disord. 2008;23 Suppl 2:S482-8. doi: 10.1002/mds.21914. PMID 18668620
- [Derived] Kim YE, Yun JY, Yang HJ, Kim HJ, Gu N, Yoon SH, Cho JY, Jeon BS. Intravenous amantadine for freezing of gait resistant to dopaminergic therapy: a randomized, double-blind, placebo-controlled, cross-over clinical trial. PLoS One. 2012;7(11):e48890. doi: 10.1371/journal.pone.0048890. Epub 2012 Nov 19. PMID 23185280